CLINICAL TRIAL: NCT00913731
Title: Quality Project to Evaluate and Validate the FAST-O Rating Scale (Fast ASessment in Acute Treatment of Psychosis-Observation)
Brief Title: Quality Project to Evaluate and Validate the FAST-O Rating Scale
Acronym: FAST-O
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: NIS-NSE-DUM-2008/1
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Acute Psychotic Symptoms
Keywords: Psychotic symptom assessments; Observational assessments of patients with acute psychotic symptoms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- psychotic patients: psychotic patients, acute ward, symptom rating scale.

SUMMARY:
The purpose of this project is to test the reliability of the FAST-O Rating Scale in patients at acute wards or psychiatric intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute psychotic symptoms attending the acute ward or psychiatric intensive care unit

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute psychotic symptoms attending the acute ward or psychiatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2009-05; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Reliability test of the FAST-O rating scale based on observational symptom ratings of patients with acute psychotic diseases | Each patients symtoms will be rated on 2 occasions, by 2-3 raters, each. First is made within 24 hrs of admission to acute psychiatric care, secondis made 14 +/- 2 days after admittance, or earlier if the patient is discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Dencker Vansvik, Study Director — Medical Department; Eva Lindström, Principal Investigator — Rättspsyk, UMAS, Malmö
Locations (5):
- Sweden (5):
  - Research Site, Helsingborg
  - Research Site, Kristianstad
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Ystad